CLINICAL TRIAL: NCT01625273
Title: Supplementation of Infant Formula With the Synbiotics (Lactobacillus Paracasei Ssp. Paracasei Strain F19 and Fructo- and Galactooligosaccharides).
Brief Title: Supplementation of Infant Formula With Synbiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arla Foods (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KB/205/2010
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Infant Formula
Keywords: F19; Lactobacillus paracasei paracasei
MeSH Terms: interventions — 11-fluoro-19-nor-dihydro-testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IF (Infant formula) (No Intervention)
- IF with L. paracasei strain F19 (Experimental)
  Interventions: Other: Lactobacillus paracasei paracasei strain F19

INTERVENTIONS:
Other: Lactobacillus paracasei paracasei strain F19 — Provided in an infant formula, 10^8 CFU per day from 28 days to 6 months of infant age
  Other Names: F19
  Arms: IF with L. paracasei strain F19

SUMMARY:
The primary hypothesis is that Lactobacillus paracasei ssp. paracasei strain F19 in an infant formula containing FOS/GOS is safe and tolerable for use in infants from 0 to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants of mothers who voluntarily resigned completely from breastfeeding
* infant age 28 days
* delivered between 38 and 42 weeks of gestation
* vaginal delivery
* birth weight > 2700 g and < 4200 g
* parent or the subject's legal representative has to speak and understand Polish

Exclusion Criteria:

* fully or partially breastfed infants
* malformations, handicaps or congenital diseases that could affect normal growth
* treatment with antibiotics
* fed infant formula with pre- and/or probiotics

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2010-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Growth (body weight, length, head circumference) | From 28 days to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hania Szajewska, MD, Principal Investigator — Samodzielny Publiczny Dziecięcy Szpital, Warsaw; Jacek Witwicki, MD, Principal Investigator — Samodzielny Publiczny Dziecięcy Szpital Kliniczny, Warsaw
Locations (1):
- Samodzielny Publiczny Dziecięcy Szpital Kliniczny, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sjodin KS, Sjodin A, Ruszczynski M, Kristensen MB, Hernell O, Szajewska H, West CE. Targeting the gut-lung axis by synbiotic feeding to infants in a randomized controlled trial. BMC Biol. 2023 Feb 20;21(1):38. doi: 10.1186/s12915-023-01531-3. PMID 36803508